CLINICAL TRIAL: NCT06596538
Title: Video-Interpreting in an Emergency Trauma Room Setting - a Feasibility Trial
Status: Withdrawn | Type: Observational
Why Stopped: Recruitment was not possible
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Christina Hafner, Principal Investigator, Medical University of Vienna
Other Study IDs: 1366/2023
Record Dates: First submitted 2023-10-25; First posted 2024-09-19 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Communication Barriers
Keywords: Communication barriers; Language barriers; Video-Interpreting; Emergency Medicine; Emergency physician

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Background: Global migration increases the likelihood of language barriers. In medical situations language barriers have a negative effect on quality of treatment and thus endanger patient safety.

In-hospital settings feasibility of video-translation has been demonstrated, yet there is lack of evidence in emergency trauma rooms. There, the physicians have to deal with time-critical decisions. Aims: This feasibility trial aims to investigate technical feasibility, usability as well as the impact on decision-making (e.g. alteration of treatment strategies). Methods: In this study 50 responsive patients with language barriers will be included. The anesthesiologic emergency physician will start video-translation via a tablet. Feasibility, quality of communication, usability as well as changes in diagnosis and treatment will be gathered and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, at least 18 years old
* awake, responsive patients
* language barrier (Albanian, Dari, Romanian, Turkish, Modern Standard Arabic, Arabic, Farsi, Russian, Hungarian, Bosnian-Croatian-Serbian, Kurdish (Kurmanci), Slovakian, Bulgarian, Polish, and Czech)

Exclusion Criteria:

* unconscious patients
* cardiac arrest patients
* delay of treatment due to e-translation
* refusal of video-translation by the patient

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: In total 50 adult patients with language barriers, who are treated in the emergency trauma room by doctors of the Department of Anaesthesia, Intensive Care Medicine and Pain Medicine will be included in this study. Inclusion and exclusion criteria as noted above will be followed.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Technical Feasibility | Directly after use of video-interpreting
  Occurance of technical problems will be reported
Usability of video-interpreting | Directly after use of video-interpreting
  The usability will be evaluated afterwards by the anesthesiologic emergency physician using a questionnaire including following items on a 7-point Likert scale (strongly disagree to strongly agree):
  * Video-interpreting was easy to use.
  * I feel comfortable to use video-interpreting during the situation.
  * The amount of time involved to use video-interpreting has been fitting for me.
  * I would use video-interpreting again.
  * Video-interpreting was useful for my healthcare practice in this situation.
Impact on emergency physician's decisions | Directly after use of video-interpreting
  The impact of video-translation will be evaluated regarding alteration of medical history or treatment (yes/no)

OTHER OUTCOMES:
Demographic parameters | Directly after use of video-interpreting
  Following characteristics of the patients will be recorded:
  Age, gender, primary diagnosis of the physician

CONTACTS AND LOCATIONS:
Locations (1):
- MUVienna, Vienna, Vienna, Austria